CLINICAL TRIAL: NCT06540989
Title: Understand Me for Life: Using Noise-augmented Automatic Speech Recognition to Improve Intelligibility in Parkinson's Disease
Brief Title: Noise-augmented Automatic Speech Recognition for Speech Treatment in Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-005
Record Dates: First submitted 2024-07-29; First posted 2024-08-07 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: One group of 42 participants with PD will be recruited and randomly assigned to either immediate treatment or deferred treatment. Twenty-one participants will receive treatment immediately after their second pre-treatment assessment. The other 21 participants will receive treatment one month after their second pre-treatment assessment. All participants will receive the same treatment.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): Participants will receive speech treatment immediately after their second pre-treatment assessment.
  Interventions: Behavioral: Immediate treatment
- Deferred treatment (Active Comparator): Participants will receive speech treatment one month after their second pre-treatment assessment. This arm receives the same speech treatment as Arm 1.
  Interventions: Behavioral: Deferred treatment

INTERVENTIONS:
Behavioral: Immediate treatment — Participants will access a web-based app using their phone to record 100 sentences every treatment session. Noise-augmented feedback will be provided to increase accuracy of speech productions.
  Arms: Immediate treatment
Behavioral: Deferred treatment — This group of participants will receive the same treatment as those in the immediate treatment group. The only difference is the timeline of treatment onset. Therefore, participants will access a web-based app using their phone to record 100 sentences every treatment session. Noise-augmented feedback will be provided to increase accuracy of speech productions.
  Arms: Deferred treatment

SUMMARY:
The goal of this clinical trial is to learn whether noise-augmented feedback using automatic speech recognition improves intelligibility and social participation in individuals with Parkinson's disease. The main questions the investigators will address are:

Does noise-augmented feedback lead to increased intelligibility, as measured by transcription accuracy scores?

Does a self-managed speech protocol lead to increased social participation, as measured by the Communicative Participation Item Bank and the Communicative Effectiveness Index questionnaires?

Participants will:

Receive 2-4 initial speech assessments in-person in our lab. Engage in speech treatment sessions at home using their phone and computer four days a week for four weeks. Four of those sessions will be directly monitored online by a speech-language pathologist. The rest of the sessions are completed by the participant.

Come to the lab for two post-treatment assessments following completion of treatment.

Come to the lab six months after treatment completion for an additional assessment.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn whether noise-augmented feedback using automatic speech recognition improves intelligibility and social participation in individuals with Parkinson's disease.

Data collection will be face-to-face at a convenient time for participants. The screening and assessment sessions will take place in the Communication, Technology, and Language Diversity Lab (Room 952a), on the 9th floor of the 528 Building at Teachers College, Columbia University (525W 120th St, New York, NY 10027).

Treatment sessions will be conducted independently by the participant in the participant's home. Four out of the 16 treatment sessions will be supervised online (via Zoom) by a licensed speech and language pathologist.

The study involves 5-7 assessment sessions (including one 6-month follow-up) and 16 treatment sessions ( = 1 month). Each participant is expected to be involved in the study for 7-8 months.

Participants will first attend a screening session to confirm eligibility, which will involve a hearing screening, a brief cognitive screening, and a brief depression screening. If the screening is successful, participants will complete two or four assessment sessions before initiation of the treatment protocol (the number of assessment sessions depends on their group allocation: immediate treatment or deferred/delayed treatment).

Screenings will only be completed once, during their first in person visit on the Teachers College campus.

In the first assessment session participants will be asked to complete voice recordings and three questionnaires. Participants will complete the same speech tasks and questionnaires in the rest of the assessment sessions. The number of assessment sessions (5 versus 7) depends on whether they are assigned to the immediate treatment group or the delayed treatment group. Group assignments are random, and participants will always receive the treatment protocol.

Each assessment session is estimated to take 60-90 minutes to complete.

Participants will complete the treatment sessions on their own using your phone and computer. Participants will be instructed to find a quiet place at home and practice their exercises at a time when they feel ok and not too tired. They will log in onto our web-based app, Understand Me for Life, to start their speech session. App instructions will be provided during the second assessment session for familiarization purposes.

Each session will contain 20 short sentences (between 3 and 7 words in length). Participants will be asked to try to complete 5 sessions in 1 hour (a total of 100 sentences), taking as many breaks as they may need. Participants will be instructed to complete 1-hour of speech exercises 4 days a week for 4 weeks. The total number of days to participate in the treatment study is 16.

ELIGIBILITY:
Inclusion Criteria:

* Participants will qualify for the study if:

  * They are 50-80 years old,
  * They have a medical diagnosis of PD,
  * They are within stages I-IV of Hoehn & Yahr Scale,
  * Their antiparkinsonian medication schedule is stable,
  * They present with mild to moderate dysarthria,
  * They score ≥ 25 in the MMSE,
  * They score ≤ 24 in the BDI-III.

Exclusion Criteria:

* Participants will be excluded from the study if they:

  * Present with atypical parkinsonism at the time of screening (or other neurological condition),
  * Underwent neurosurgery treatment (DBS),
  * Received intensive voice-focused treatment less than three months prior to their involvement in the current study,
  * Present with any speech or voice pathology that is unrelated to PD.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Intelligibility | 3 years
  Transcription accuracy (% words correctly understood by listeners)

SECONDARY OUTCOMES:
Social participation | 7-8 months
  Communicative Participation Item Bank questionnaire (10 questions, 0 = very much to 3 = not at all)
Social participation | 7-8 months
  Communication Effectiveness Index questionnaire (8 questions, 1 = not at all effective, 4 = very effective)

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Moya-Galé, Ph.D., Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No